CLINICAL TRIAL: NCT00824174
Title: Body Image Functioning Among Surgically Treated Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0080
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Head and Neck Cancer; Skin Cancer
Keywords: Questionnaire; Head and Neck Cancer; Skin Cancer; Body Image; Surgical Treatment; Oral Cavity Cancer; Cutaneous Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Skin Neoplasms; Mouth Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire: 1 questionnaire, about 15-20 minutes.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 1 questionnaire, about 15-20 minutes.
  Other Names: Survey

SUMMARY:
Objectives:

The purpose of this study is to obtain descriptive information about the nature and extent of body image concerns among surgical patients with head and neck cancer, satisfaction with care received regarding body image issues, and interest in psychosocial services targeting body image disturbance. Findings from this study provide important preliminary data to guide future large scale research on the critical, yet understudied, psychosocial issue of body image functioning for head and neck cancer patients. Information obtained from this study can specifically be used to facilitate the development of appropriate disease-specific body image instruments and to determine the need for body image focused psychosocial interventions to enhance quality of life and the survivorship experience for these patients.

Primary Aims

1. To characterize the nature and extent of body image concerns in surgically treated patients with head and neck cancer and determine preferences for psychosocial intervention.
2. To compare body image and quality of life outcomes for patients at different time points relative to initiation of treatment. Specific time points of interest are pre-treatment, within one year of initial surgical treatment, and greater than 1 year following initial surgical treatment.

Secondary Aim

1. To compare body image and quality of life outcomes for patients with oral cavity, cutaneous, and midface cancers.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to fill out 1 questionnaire. This questionnaire can be filled out while you are waiting to be seen by your head and neck doctor and will take about 15-20 minutes to complete.

In this questionnaire, you will be asked questions such as your age, gender, education level, and smoking history. You will also be asked about your treatment for cancer and how it has affected your appearance and body. There will also be questions about your mood, physical health, alcohol use, and social well-being.

Length of Study:

You will be off study after you complete the questionnaire.

This is an investigational study. Up to 350 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Able to provide written informed consent to participate
3. Diagnosis of oral cavity, cutaneous or other midface cancer involving the head and neck region
4. Treatment plan includes surgical intervention
5. English speaking

Exclusion Criteria:

1. Significant preexisting facial disfigurement from a previous trauma or congenital defect
2. Diagnosis of a serious mental illness involving formal thought disorder (e.g., schizophrenia) documented in medical record
3. Cognitive impairment (e.g., dementia, delirium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, 18 years or older, with oral cavity or cutaneous cancer receiving surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2008-12; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Body image outcomes (i.e., Body Image Scale) for patients at different time points relative to initiation of treatment | Specific time points of interest are pre-treatment, within one year of initial surgical treatment, and greater than 1 year following initial surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Fingeret, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org